CLINICAL TRIAL: NCT02372656
Title: Comparison Of Efficacy Of Locally Delivered 1.2% Simvastatin And 1% Metformin Gel In Chronic Periodontitis: A Randomized Placebo Controlled Clinical Trial
Brief Title: Simvastatin and Metformin in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/10C/2013-14
Record Dates: First submitted 2014-11-30; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Periodontitis
Keywords: Simvastatin, Metformin, Chronic periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Metformin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Group (Placebo Comparator): Placebo gel without active ingredient to be delivered at baseline, 3, 6 and 9 months.
  Interventions: Drug: Placebo gel
- 1% Metformin (Active Comparator): 1% metformin gel to be delivered at baseline, 3, 6 and 9 months.
  Interventions: Drug: 1% Metformin
- 1.2% Simvastatin (Active Comparator): 1.2% Simvastatin to be delivered at baseline, 3, 6 and 9 months.
  Interventions: Drug: 1.2% Simvastatin

INTERVENTIONS:
Drug: Placebo gel — Placebo gel to be delivered in intrabony sites of chronic periodontitis subjects at baseline, 3,6 and 9 months.
  Other Names: Placebo group
  Arms: Placebo Group
Drug: 1% Metformin — 1% Metformin gel to be delivered in intrabony sites of chronic periodontitis subjects at baseline, 3,6 and 9 months.
  Other Names: 1% Metformin group
  Arms: 1% Metformin
Drug: 1.2% Simvastatin — 1.2% Simvastatin gel to be delivered in intrabony sites of chronic periodontitis subjects at baseline, 3,6 and 9 months.
  Other Names: 1.2% Simvastatin group
  Arms: 1.2% Simvastatin

SUMMARY:
This randomized controlled clinical trial compares efficacy of 1.2% simvastatin with 1% metformin in chronic periodontitis subjects.

DETAILED DESCRIPTION:
Aim: To compare the efficacy of locally delivered 1.2% SMV gel and 1% MF gel in treatment of intrabony defects in chronic periodontitis subjects and compare it with placebo gel.

Methods: Ninety subjects were categorized into three treatment groups: 1.2% Simvastatin (SMV), 1% Metformin (MF) and placebo gel after Scaling and root planning (SRP). Clinical parameters were recorded at baseline, 3, 6 and 9 months; they included plaque index (PI), modified sulcus bleeding index (mSBI), pocket probing depth (PPD), and clinical attachment level (CAL). Radiologic assessment of intra bony defect (IBD) and percentage defect depth reduction (DDR%) was done at baseline, 6 months and 9 months interval using computer-aided software

Results: Mean PPD reduction and mean CAL gain was found to greater in SMV group than MF and placebo group at all visits. The DDR% was greater in SMV group as compared to MF and placebo group.

Conclusion: There was greater decrease in mSBI and PPD and more CAL gain with significant IBD depth reduction at the sites treated with SMV and MF as an adjunct to SRP in chronic periodontitis subjects with intrabony defects as compared to placebo. The effect was greater in case of SMV group, however there was no significant defect depth reduction as compared to MF.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy subjects
* Pocket depth ≥ 5 mm
* Clinical attachment level ≥ 4 mm and vertical bone loss ≥ 3 mm on intraoral periapical radiographs, with no history of periodontal therapy in the last 6 months

Exclusion Criteria:

* Subjects allergic to MF or SMV
* Those on systemic MF or SMV therapy
* Subjects with aggressive periodontitis
* Immunocompromised subjects
* Use of tobacco in any form, alcoholics
* Lactating and pregnant females

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in defect depth reduction from baseline to 6 months and from baseline to 9 months | Baseline to 6 months and Baseline to 9 months
  Radiographic defect depth reduction to measured at baseline, 6 and 9 months interval.

SECONDARY OUTCOMES:
Plaque index will be measured at 3, 6 and 9 months | 3,6 and 9 months
Modified sulcular bleeding index at 3, 6 and 9 months | 3 , 6 and 9 months
Probing pocket depth at 3, 6 and 9 months | 3 , 6 and 9 months
Clinical attachment level at 3, 6 and 9 months | 3 , 6 and 9 months